CLINICAL TRIAL: NCT04012255
Title: A Trial to Demonstrate Bioequivalence Between Semaglutide Formulations With the DV3396 Pen-injector and With the PDS290 Pen-injector in Subjects With Overweight or Obesity
Brief Title: A Research Study to Compare Two Forms of Semaglutide in Two Different Pen-injectors in People With Overweight or Obesity
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial was terminated for strategic reasons.
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9536-4475; U1111-1221-9644 (Other: World Health Organization (WHO)); 2018-003923-13 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2019-07-05; First posted 2019-07-09 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DV3396 (Experimental): Participants will receive once-weekly doses of semaglutide administered with the DV3396 pen-injector (test drug product)
  Interventions: Drug: Semaglutide (administered by DV3396 pen)
- PDS290 (Active Comparator): Participants will receive once-weekly doses of semaglutide administered with the PDS290 pen-injector (comparator drug product)
  Interventions: Drug: Semaglutide (administered by PDS290 pen)

INTERVENTIONS:
Drug: Semaglutide (administered by DV3396 pen) — Increasing doses of semaglutide given subcutaneously (sc, under the skin) in the stomach for 21 weeks
  Arms: DV3396
Drug: Semaglutide (administered by PDS290 pen) — Increasing doses of semaglutide given sc in the stomach for 21 weeks
  Arms: PDS290

SUMMARY:
The study will look at how two different forms of semaglutide reach and stay in the blood after injection. None of the two forms of semaglutide have been approved by the authorities to treat obesity. Participants will get 1 of the 2 forms of semaglutide - which one is decided by chance. Participants will get the medicine as an injection under the skin of the stomach with the use of a pen-injector. The type of pen-injector is different for the two forms of semaglutide. The study staff will teach participants how to inject themselves with the medicine. As part of this training participants will self inject placebo (dummy medication) 3 times. Participants will take an injection once a week and will get 21 injections in total of study medication. The study will last for about 27-30 weeks. Participants will have 25 study visits with the study doctor. For 2 of the visits, participants will stay in the clinic for 3 days and 2 nights. Participants may have to stop the study if the study doctor thinks that there are risks for their health. Women cannot take part if they are pregnant, breast-feeding or planning to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-65 years (both inclusive) at the time of signing informed consent
* Body mass index (BMI) between 27.0 and 34.9 kg/m^2 (both inclusive)
* Body weight between 70.0 and 130.0 kg (both inclusive)

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using a highly effective contraceptive method
* Any disorder which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol
* Inability or unwillingness to perform self-injection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-10-22 (Actual)

PRIMARY OUTCOMES:
AUC0-168h,2.4mg,SS: Area under the semaglutide concentration time curve following the last administration of semaglutide s.c. 2.4 mg | 0-168 hours (Day 141-148) after last 2.4 mg dose
  h*nmol/L
Cmax,2.4mg,SS: Maximum observed semaglutide concentration following the last administration of semaglutide s.c. 2.4 mg | 0-168 hours (Day 141-148) after last 2.4 mg dose
  nmol/L

SECONDARY OUTCOMES:
AUC0-168h,1mg,SS: Area under the semaglutide concentration time curve following the last administration of semaglutide s.c. 1 mg | 0-168 hours (Day 78-85) after last 1 mg dose
  h*nmol/L
Cmax,1mg,SS: Maximum observed semaglutide concentration following the last administration of semaglutide s.c. 1 mg | 0-168 hours (Day 78-85) after last 1 mg dose
  nmol/L
Tmax,2.4mg,SS: Time of maximum observed semaglutide concentration after last 2.4 mg dose | 0-168 hours (Day 141-148) after last 2.4 mg dose
  h
Tmax,1mg,SS: Time of maximum observed semaglutide concentration after last 1 mg dose | 0-168 hours (Day 78-85) after last 1 mg dose
  h
t½: Terminal elimination half-life of semaglutide after last 2.4 mg dose | 0-1176 hours (Day 141-190) after last 2.4 mg dose
  h
Cl/F2.4mg: Total apparent clearance of semaglutide after last 2.4 mg dose | 0-168 hours (Day 141-148) after last 2.4 mg dose
  L/h
Cl/F1mg: Total apparent clearance of semaglutide after last 1 mg dose | 0-168 hours (Day 78-85) after last 1 mg dose
  L/h
Vss/F2.4mg: Apparent volume of distribution at steady-state of semaglutide after last 2.4 mg dose | 0-168 hours (Day 141-148) after last 2.4 mg dose
  L
Vss/F1mg: Apparent volume of distribution at steady-state of semaglutide after last 1 mg dose | 0-168 hours (Day 78-85) after last 1 mg dose
  L
Change in body weight | From baseline (Day 1, pre-dose) until the end of treatment (Day 148)
  percent

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (2):
- Germany (2):
  - Novo Nordisk Investigational Site, Mainz
  - Novo Nordisk Investigational Site, Neuss

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com